CLINICAL TRIAL: NCT04138888
Title: Single Dose Crossover Comparative Bioavailability Study of Olmesartan Medoxomil/Hydrochlorothiazide 40 mg/25 mg Film-Coated Tablets in Healthy Adult Subjects / Fasting State
Brief Title: A Bioequivalence Study of Two Different Formulations of Olmesartan Medoxomil/ Hydrochlorothiazide After a Single Oral Dose Administration Under Fasting Conditions
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Altasciences Company Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: PTL-P0-847
Record Dates: First submitted 2019-10-23; First posted 2019-10-25 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-10

CONDITIONS: Bioequivalence
Keywords: Olmesartan medoxomil/hydrochlorothiazide; Bioequivalence; Olmetec Plus®
MeSH Terms: interventions — Olmesartan Medoxomil; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The randomization code will not be available to the personnel of the bioanalytical facility until the bioanalytical tables have been finalized and audited by the Quality Assurance (QA) department. Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence AB (Other): 16 subjects assigned to the sequence AB will receive a single 40 mg/25 mg dose of the test product Olmesartan Medoxomil/ Hydrochlorothiazide (1 x 40 mg/ 25 mg tablet), marked as A in the sequence, in Period 1 and a single 40 mg/25 mg dose of the reference product Olmetec® Plus (1 x 40 mg/ 25 mg tablet), marked as B in the sequence, in period 2. These treatments will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Olmesartan Medoxomil/Hydrochlorothiazide 40 Mg/25 Mg film-coated tablets for oral use; Drug: Olmetec® Plus 40 Mg/25 Mg film-coated tablets for oral use
- Sequence BA (Other): 16 subjects assigned to the sequence BA will receive a single 40 mg/25 mg dose of the reference product Olmetec® Plus (1 x 40 mg/ 25 mg tablet), marked as B in the sequence, in Period 1 and a single 40 mg/25 mg dose of the test product Olmesartan Medoxomil/ Hydrochlorothiazide (1 x 40 mg/ 25 mg tablet), marked as A in the sequence, in period 2. These treatments will be administered orally with approximately 240 mL of water, in the morning, following a 10-hour overnight fast. The tablet must be swallowed whole and must not be chewed or broken.
  Interventions: Drug: Olmesartan Medoxomil/Hydrochlorothiazide 40 Mg/25 Mg film-coated tablets for oral use; Drug: Olmetec® Plus 40 Mg/25 Mg film-coated tablets for oral use

INTERVENTIONS:
Drug: Olmesartan Medoxomil/Hydrochlorothiazide 40 Mg/25 Mg film-coated tablets for oral use — Olmesartan Medoxomil/Hydrochlorothiazide is manufactured by Pharmtechnology LLC, Republic of Belarus. Each tablet contains 40 mg of olmesartan medoxomil and 25 mg of hydrochlorothiazide.
  Other Names: The test product
Drug: Olmetec® Plus 40 Mg/25 Mg film-coated tablets for oral use — Olmetec® Plus is manufactured by Daiichi Sankyo Europe GmbH, Germany. Each tablet contains 40 mg of olmesartan medoxomil and 25 mg of hydrochlorothiazide.
  Other Names: The reference product

SUMMARY:
This single dose study was designed in accordance with EMA (the European Medicines Agency) regulatory guidelines, with the aim of characterizing the bioavailability of olmesartan medoxomil/ hydrochlorothiazide in the two formulations (Olmesartan Medoxomil/ Hydrochlorothiazide (HCTZ), 40 mg/ 25 mg film-coated tablets (Manufacturer: Pharmtechnology LLC, Republic of Belarus) and Olmetec Plus® (Olmesartan Medoxomil/ Hydrochlorothiazide), 40 mg/25 mg film-coated tablets, (Manufacturer: Daiichi Sankyo Europe GmbH, Germany)) in healthy subjects. As this is a bioequivalence trial where each subject received each study treatment in a crossover fashion, a control group was not included. Within the clinical portion of the study each subject received a single oral dose of the test and the reference formulation in compliance with the generated randomization code. The primary study endpoints were the pharmacokinetic (PK) parameters Cmax and AUC0-t of olmesartan and hydrochlorothiazide.

DETAILED DESCRIPTION:
This is a single center, randomized, single dose, laboratory-blinded, 2-period, 2-sequence, crossover study design, in which 32 healthy adult subjects received one of the study treatments during each study period.

The objective of this study is to determine the bioequivalence of two different formulations of olmesartan medoxomil/ HCTZ after a single oral dose administration under fasting conditions.

The intra-subject variation following a single dose of olmesartan/ HCTZ appears to be around 25% for Cmax and around 18% for AUC0-T for olmesartan and around 18% for Cmax and around 13% for AUC0-T for HCTZ. Statistically, given that the expected Test to Reference ratio of geometric LSmeans should fall within 95 and 105%, it is estimated that the lowest number of subjects to meet the 80 to 125% bioequivalence range for each analyte with a statistical a priori power of at least 80% is about 28.

Therefore, the inclusion of 32 subjects should be sufficient to account for the possibility of drop-outs, variations around the estimated intra-subject CV and to conclude in favor of the hypothesis of bioequivalence with sufficient statistical power. A Caucasian population will be enrolled to minimize variability and optimize detection of differences between the Test and Reference formulations without regard to race.

Subject eligibility for this study will be determined at the screening visit and eligible subjects will be admitted to the clinical research unit at least 10 hours prior to drug administration for each study period.

Standbys should be recruited and available to replace any subject who withdraws prior to the first drug administration.

On-study drop-outs will not be replaced. Altasciences will generate the randomization code with a computer program according to the study design, the number of subjects and the sequence of treatment administration. The random allocation of each sequence of treatment administration to each subject will be done in such a way that the study is balanced. Once generated, the randomization code will be final and will not be modified. Eligible subjects will be randomized to one of two treatment sequences. There will be two sequences in the study: AB and BA, where A = the test product, B = the reference product (see detailed description of A and B items in Section "Arms and Interventions").

For each study period, subjects will receive a single 40 mg/25 mg oral dose of olmesartan medoxomil/HCTZ, under fasting conditions and undergo a 48-hour PK sample collection. Study participants will be aware they will receive different formulations of the same drug, without being informed which product (Test or Reference) is being administered. The date and time of each dose will be recorded. For each subject, all scheduled postdose activities and assessments will be performed relative to the time of study drug administration.

Subjects will fast overnight (no food or drink except water), for a minimum of 10 hours prior to dosing. Fasting will continue for at least 4 hours following drug administration, after which a standardized lunch will be served. A supper and a light snack will be served at appropriate times thereafter, but not before 9 hours after dosing.

Water will be provided as needed until 1 hour predose. Water will be allowed beginning 1 hour after the administration of the drug.

A total of 42 blood samples will be collected (1 tube of 3 mL for olmesartan and 1 tube of 3 mL for HCTZ at each time point) in each study period for PK assessments. The first blood sample will be collected prior to drug administration while the others will be collected up to 48 hours after drug administration.

Given that olmesartan medoxomil is rapidly and completely converted to the pharmacologically active metabolite, olmesartan, and that no intact olmesartan medoxomil or intact side chain medoxomil moiety have been detected in plasma1,2, olmesartan medoxomil cannot be reliably measured. Therefore, the analytes to be measured in the study will be olmesartan and hydrochlorothiazide. Olmesatran and HCTZ plasma concentrations will be measured according to validated bioanalytical methods.

Subjects are to be discharged from the clinic after the 24-hour postdose PK sample collection, and following medical approval. However, they may be advised to stay at the clinical site for safety reasons, if judged necessary by the physician in charge. Subjects will return to the clinic for blood collections at 48 hours postdose.

The expected terminal half-life values observed after a single oral 40 mg/25 mg dose of olmesartan medoxomil/HCTZ film-coated tablet under fasting conditions are 8.6 hours for olmesartan and 10.3 hours for HCTZ. To avoid any carry-over effect, a wash-out of 7 calendar days is planned between drug administrations, corresponding to more than 16 times the expected half-life of the moieties to be measured. The decision of which subjects will be included in the PK analysis is to be documented by the pharmacokineticist (or delegate) and approved by the sponsor before the start of the sample analysis by the bioanalytical facility.

Subjects who are expected to provide evaluable PK data for both the Test and Reference products (based on viable PK samples) will be included in the pharmacokinetic analysis.

Concentration data of the remaining subjects will be presented separately. Subjects who do not complete the sampling schedule of one or more study periods may be included in the PK and statistical analysis and bioequivalence determination for only the PK parameters that are judged not to be affected by the missing sample(s).

Statistical analysis of Tmax will be based on a non-parametric approach. Statistical analysis of all other PK parameters will be based on an Analysis of Variance (ANOVA) model. Two-sided 90% confidence interval of the ratio of geometric Least-Square means (LSmeans) obtained from the ln transformed PK parameters will be calculated.

Statistical inference of olmesartan and HCTZ will be based on a bioequivalence approach using the following standards: the ratio of geometric LSmeans with corresponding 90% confidence interval calculated from the exponential of the difference between the Test and the Reference for the ln-transformed parameters Cmax and AUC0-T should all be within the 80.00 to 125.00% bioequivalence range.

The safety population will include all subjects who received at least one dose of one of the IPs. Safety assessments will include vital signs, clinical laboratory tests, and AE monitoring. Additional safety measurements may be performed at the discretion of the investigator for reasons related to subject safety. The physician in charge will be present at the clinical site for at least the first 4 hours following each drug administration and will remain available at all times throughout the study.

Total study duration: up to 38 days (including screening).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form (ICF);
2. Stated willingness to comply with all study procedures and availability for the duration of the study;
3. Healthy Caucasian adult male or female;
4. If female, meets one of the following criteria:

   A. Physiological postmenopausal status, defined as the following:
   1. absence of menses for at least one year prior to the first study drug administration (without an alternative medical condition); and
   2. Follicle stimulating hormone (FSH) levels ≥40 mIU/mL at screening; or

   B. Surgical postmenopausal status, defined as the following:
   1. bilateral oophorectomy; and
   2. absence of menses for at least 90 days prior to the first study drug administration; and
   3. FSH levels ≥ 40 mIU/mL at screening; or C. Hysterectomy with FSH levels ≥ 40 mIU/mL at screening. If the postmenopausal subject has an FSH of < 40 mIU/mL, but meets the above criteria in either (A), (B) or (C) and all the other inclusion criteria, the subject may be included in the study if the estradiol serum level measured at screening is equal to or below 150 pmol/L;
5. Aged at least 18 years but not older than 50 years;
6. Body mass index (BMI) within 18.50 kg/m2 to 30.00 kg/m2, inclusively;
7. Non- or ex smoker (An ex smoker is defined as someone who completely stopped using nicotine products for at least 180 days prior to the first study drug administration);
8. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without clinical significance, as determined by an investigator;
9. Have no clinically significant (CS) diseases captured in the medical history or evidence of CS findings on the physical examination (including vital signs) and/or electrocardiogram (ECG), as determined by an investigator.

Exclusion Criteria:

1. Female who is lactating at screening;
2. Female who is pregnant according to the pregnancy test at screening;
3. Seated pulse rate less than 50 beats per minute (bpm) or more than 100 bpm at the screening visit and prior to the first study drug administration;
4. Seated blood pressure below 110/60 mmHg at the screening visit and prior to the first study drug administration;
5. History of significant hypersensitivity to olmesartan and HCTZ or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs;
6. Presence or history of significant gastrointestinal, liver or kidney disease, or any other condition that is known to interfere with drug absorption, distribution, metabolism or excretion, or known to potentiate or predispose to undesired effects;
7. History of significant cardiovascular, pulmonary, hematologic, neurological, psychiatric, endocrine, immunologic or dermatologic disease;
8. Presence of CS ECG abnormalities at the screening visit, as defined by medical judgment;
9. History of rare hereditary problems of galactose and/or lactose intolerance, lactase deficiency or glucose-galactose malabsorption;
10. Maintenance therapy with any drug or significant history of drug dependency or alcohol abuse (> 3 units of alcohol per day [1 unit = 10 mL of pure alcohol], intake of excessive alcohol, acute or chronic);
11. Any CS illness in the 28 days prior to the first study drug administration;
12. Use of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) in the 28 days prior to the first study drug administration, that in the opinion of an investigator would put into question the status of the participant as healthy;
13. Any history of tuberculosis;
14. Positive test result for alcohol and/or drugs of abuse at screening or prior to the first drug administration;
15. Positive screening results to HIV Ag/Ab combo, hepatitis B surface antigen or hepatitis C virus tests;
16. Inclusion in a previous group for this clinical study;
17. Intake of olmesartan medoxomil or HCTZ in the 28 days prior to the first study drug administration;
18. Intake of an Investigational Product (IP) in the 28 days prior to the first study drug administration;
19. Donation of 50 mL or more of blood in the 28 days prior to the first study drug administration;
20. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the 56 days prior to the first study drug administration.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-10-31 (Actual); Primary Completion 2019-12-24 (Estimated); Study Completion 2019-12-24 (Estimated)

PRIMARY OUTCOMES:
Cmax of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Maximum observed concentration in plasma
AUC0-t of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Cumulative area under the concentration time curve calculated from 0 to TLQC using the linear trapezoidal method, where TLQC represents time of last observed quantifiable concentration

SECONDARY OUTCOMES:
Tmax of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Time of maximum observed concentration; if it occurs at more than one time point, Tmax is defined as the first time point with this value
TLQC of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Time of last observed quantifiable concentration
AUC0-∞ of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Area under the concentration time curve extrapolated to infinity, calculated as AUC0-T + ĈLQC/λZ, where ĈLQC is the predicted concentration at time TLQC
Residual area of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Extrapolated area (i.e. percentage of AUC0-∞ due to extrapolation from TLQC to infinity).
Time point where the log-linear elimination phase begins (TLIN) of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Lower limit on time for values included in the calculation of λz
λZ of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Apparent elimination rate constant, estimated by linear regression of the terminal linear portion of the log concentration versus time curve
Terminal elimination half-life (Thalf) of olmesartan and HCTZ in plasma after administration of the test and the reference products. | Time points 0.00 (prior to each drug administration) and 0.33, 0.67, 1.00, 1.33, 1.67, 2.00, 2.33, 2.67, 3.00, 3.33, 3.67, 4.00, 4.50, 5.00, 6.00, 8.00, 10.00, 12.00, 24.00, 48.00 hours after each drug administration.
  Terminal elimination half-life, calculated as ln(2)/λZ
Number of treatment-emergent adverse events for the test and the reference products. | Up to 11 days (after the first drug administration until the end of the period of 1 day following the last blood sample of the study)
  The safety population will include all subjects who received at least one dose of the test or the reference product. Any significant changes will be recorded as treatment-emergent adverse events only if they are judged clinically significant by the qualified investigator or delegate.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, MD, Principal Investigator — Altasciences Company Inc.
Locations (1):
- Altasciences Company Inc., Mount Royal, Quebec, Canada